CLINICAL TRIAL: NCT04969575
Title: Exploring Single Step Culture Medium Refreshment Effect on Embryo Ploidy Rate: A Benchtop Incubator Prospective Study
Brief Title: A Benchtop Incubator Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Ibrahim Elkhatib, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2105-ABU-008-IK
Record Dates: First submitted 2021-07-11; First posted 2021-07-20 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Infertility
Keywords: IVF; incubator; aneuploidy; embryoscope; embryo; ICSI
MeSH Terms: conditions — Infertility; Aneuploidy | interventions — Insemination; Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- day 3 refreshment: All MII oocytes will be inseminated by ICSI 39-41 hours post final oocyte maturation trigger.
  Following ICSI, oocytes will be cultured in 2-4 culture dishes placed in 2 separate chambers.
  Media refreshment: Zygote scoring on day 1 (18-20hpi). Culture medium refreshment will be done 67-69 hours post insemination (Day3). Embryo grading will not be done day2-5. Culture media preparation and refreshment: 30µL of culture medium (Global total LP is added to each well of the 8 wells of LifeGlobal GPS Dish (EGPS-010) and 50µL to the center 3 drops.
  Dishes will be equilibrated overnight in a CO2 incubator. Embryo grading should be done prior to media refreshment. Time out of the incubator during media refreshment will be assessed on day 3 and day 5.
  One operator should perform the ICSI. In case of multiple operators, each operator's injected oocytes will be split between the 2 groups.
  Interventions: Other: Insemination and culture; Other: Media refreshment Group 1; Other: Culture media preparation and refreshment; Other: Embryo grading
- day 5 refreshment: All MII oocytes will be inseminated by ICSI 39-41 hours post final oocyte maturation trigger.
  Following ICSI, oocytes will be cultured in 2-4 culture dishes placed in 2 separate chambers.
  Media refreshment and embryo grading timings: Zygote scoring on day 1 (18-20hpi). Embryo grading and culture media refreshment will be done 114-118 hours post insemination (Day5).
  Culture media preparation and refreshment: 30µL of culture medium (Global total LP is added to each well of the 8 wells of LifeGlobal GPS Dish (EGPS-010) and 50µL to the center 3 drops. Dishes will be equilibrated overnight in a CO2 incubator.
  Embryo grading and media refreshment is done prior to blastocyst biopsy. Time out of the incubator during media refreshment will be assessed on day 3 and day 5.
  One operator should perform the ICSI. In case of multiple operators, each operator's injected oocytes will be split between the 2 groups.
  Interventions: Other: Insemination and culture; Other: Culture media preparation and refreshment; Other: Embryo grading; Other: Media refreshment Group 2

INTERVENTIONS:
Other: Insemination and culture — All MII oocytes will be inseminated by ICSI 39-41 hours post final oocyte maturation trigger.
Other: Media refreshment Group 1 — Zygote scoring on day 1 (18-20hpi). Culture medium refreshment will be done 67-69 hours post insemination (Day3).
  Groups: day 3 refreshment
Other: Culture media preparation and refreshment — 30µL of culture medium (Global total LP is added to each well of the 8 wells of LifeGlobal GPS Dish (EGPS-010) and 50µL to the center 3 drops.
  Dishes will be equilibrated overnight in a CO2 incubator.
Other: Embryo grading — Should be done prior to media refreshment. For group 2, embryo grading and media refreshment is done prior to blastocyst biopsy.
Other: Media refreshment Group 2 — Zygote scoring on day 1 (18-20hpi). Culture media refreshment will be done 114-118 hours post insemination (Day5).
  Groups: day 5 refreshment

SUMMARY:
The use of extended embryo culture to the blastocyst stage and preimplantation genetic testing for aneuploidy (PGT-A) has enabled identification and selection of embryos with the best developmental potential and improved in vitro fertilization (IVF) clinical outcomes. While numerous types of commercially available human embryo culture media exist for culture to the blastocyst stage, the impact of culture conditions on blastocyst development and aneuploidy formation is not well understood.

Culture conditions are very important for the success of the IVF cycle, many of the factors involved in the process have been extensively studied, including the use of sequential culture medium vs single step culture medium, humidified incubators vs dry incubators and refreshing the medium on day 3 vs uninterrupted culture till day 5. However, none of the studies investigated the effect on euploid rate in a sibling oocyte design with PGT-A, which requires culture till day 7.

DETAILED DESCRIPTION:
It is considered a routine practice to grade the embryos on day 3 of development, which will require disturbing the culture conditions by annotating the embryos using inverted microscopes. Extended culture to day 7 is required in order to perform trophectoderm biopsy required for PGT-A. There are several culture factors that can affect embryo development, such as the pH, which is controlled through the concentration of CO2, and also the osmolality, which is the concentration of solute per liter of solution. Evaporation of the solution due to the exposure to high temperature (37°C) can change the concentrations and hence compromise embryo development.

To reduce the rate of evaporation, culture droplets are covered with a layer of mineral oil. Humidified incubators can also reduce the rate of evaporation. However, in the case of dry incubators, such as benchtop incubators, replenishing the culture medium at least once -by moving the embryos to a new culture dish- during these 7 days of culture might be the solution.

Since single-step medium is designed to sustain embryo development for 5 continuous culture days, while some laboratories culture embryos for 7 days, refreshing the culture medium is inevitable either on day 3 or day 5 of development.

There is no concrete evidence on which of these practices will provide a better environment for embryo development. Moreover, none of the studies investigated the effect of single-step culture medium changeover on day 3 or day 5, on the chromosomal errors (aneuploidy/mosaicism). Investigators aim in this prospective sibling oocyte study, to explore which day of culture medium refreshment (day 3 or day 5) provides a higher rate of euploid blastocysts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a minimum of 8 - 10 follicles during ovarian stimulation
* Patients with a minimum of 8 mature oocytes
* PGT-A
* ICSI
* BMI<35
* Age 18- 40
* Fresh or frozen ejaculated sperm >10,000 motile sperm
* Any ovarian stimulation
* Embryos cultured in benchtop incubator

Exclusion Criteria:

* PGT-M or PGT-SR
* Previous history of embryo arrest
* Endometriosis
* History of previous treatment which may impact the ovarian reserve (adnexal surgery, chemotherapy, radiation…)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The study is eligible to all patients, meeting the inclusion criteria, undergoing a fertility treatment with PGT-A analysis at the blastocyst stage
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Blastocyst ploidy | 3 days
  determined after biopsy of trophectoderm cells, taken from the blastocyst on day 5, 6 or 7 from development

SECONDARY OUTCOMES:
Cycle ploidy rate | 1 day
  the number of euploid embryos in the group divided by the total number of 2PN (both groups)
Mosaicism Frequency | 1 day
  defined as the rate of mosaic errors in aneuploid embryos. This includes full mosaic embryos or aneuploid embryos with 1 or more mosaic chromosome aberration
Blastocyst quality at time of biopsy | 1 day
  Four Embryo Quality Scores (EQ1, 2, 3, 4) based on the expansion stage of the blastocyst, the grade of the inner cell mass and the grade of the trophectoderm.
Blastulation rate | 5 days
  ability of the embryo to form a cavity (=to blastulate) 114-118 hours post ICSI. Number of blastocysts divided by the number of 2PN

CONTACTS AND LOCATIONS:
Overall Officials: IBRAHIM ELKHATIB, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Bavister BD, Poole KA. Duration and temperature of culture medium equilibration affect frequency of blastocyst development. Reprod Biomed Online. 2005 Jan;10(1):124-9. doi: 10.1016/s1472-6483(10)60813-9. PMID 15705308
- [Background] Costa-Borges N, Belles M, Meseguer M, Galliano D, Ballesteros A, Calderon G. Blastocyst development in single medium with or without renewal on day 3: a prospective cohort study on sibling donor oocytes in a time-lapse incubator. Fertil Steril. 2016 Mar;105(3):707-713. doi: 10.1016/j.fertnstert.2015.11.038. Epub 2015 Dec 12. PMID 26690010
- [Background] Pena F, Davalos R, Rechkemmer A, Ascenzo A, Gonzales M. Embryo development until blastocyst stage with and without renewal of single medium on day 3. JBRA Assist Reprod. 2018 Mar 1;22(1):49-51. doi: 10.5935/1518-0557.20180012. PMID 29318868
- [Background] Krasnopolskaya KV, Beketova AN, Sesina NI, capital ES, Cyrillichinchenko NK, Badalyan GV, Sudarikova NM, Bocharova TV, Zakharchenko EO. The effect of short-term disturbance of day 3 embryo culture on the development and implantation. Gynecol Endocrinol. 2019;35(sup1):1-4. doi: 10.1080/09513590.2019.1632083. PMID 31532309
- See also: 1. Mori, C., Kuwayama, M., Silber, S., Kagawa, N., Kato, H. Water evaporation and osmolality change of human embryo culture media in humid or in dry culture systems. Fertil. Steril. 2010; 94: s151 — https://doi.org/10.1016/j.fertnstert.2010.07.607